CLINICAL TRIAL: NCT03926312
Title: Smart Device-based Cardiac Rehabilitation After Myocardial Intervention
Acronym: SmartRehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Peter Wohlfahrt, Principal Investigator, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SmartRehab
Record Dates: First submitted 2019-04-21; First posted 2019-04-24 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; cardiac rehabilitation; smart device; remote monitoring; telemonitoring; low physical activity; risk factors control
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart device-based rehabilitation (Experimental): One month after myocardial infarction, patients will receive a smart band and a cellphone in order to transmit data on physical activity to electronic health record. A study nurse will periodically check compliance with recommended physical activity and intervene in the case of non-compliance.
  Interventions: Device: Smart device-based cardiac rehabilitation
- Control group (No Intervention): Patients will receive a guideline directed recommendation to increase physical activity to 30 minutes of moderate physical activity a week.

INTERVENTIONS:
Device: Smart device-based cardiac rehabilitation — A smart device coupled with remote monitoring will be used to increase physical activity of patients after myocardial infarction with a history of low physical activity.
  Arms: Smart device-based rehabilitation

SUMMARY:
The aim of this study is to evaluate the influence of cardiac rehabilitation based on smart band use and telemonitoring on functional capacity change and risk factors control among patients hospitalized for acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent with the study
2. Men and women >18 years of age
3. Patients ≥1 and ≤6 months after type I myocardial infarction
4. Physical inactivity before MI defined as the absence of moderate to vigorous exercise for at least 30 minutes 5 or more days a week

Exclusion Criteria:

1. Heart failure NYHA IIIB-IV
2. Planned coronary revascularization
3. Planned major surgery within the next 12 months
4. Inability to walk for any reason
5. Comorbidities that would preclude adherence to the rehabilitation program (e.g. arthrosis, active malignancy, major depression or other significant psychiatric disorder, cognitive impairment) - at the discretion of the physician
6. Life expectancy less than 12 months
7. Pregnancy
8. Inability to operate the smart-watch

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Functional capacity change | 3 months
  6-minute walk test distance and maximal oxygen consumption (VO2 max) change after 3 months of the intervention

SECONDARY OUTCOMES:
Waist circumference | 3 months
  Waist circumference change after 3 months of the intervention
Body fat percentage | 3 months
  Body fat percentage change after 3 months of the intervention
Smoking cessation | 3 months
  Smoking cessation after 3 months of the intervention
Lipid levels | 3 months
  Lipid levels change after 3 months of the intervention
Blood pressure | 3 months
  Blood pressure change after 3 months of the intervention
Glycated hemoglobin | 3 months
  Glycated hemoglobin change after 3 months of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wohlfahrt, MD, PhD, Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, CZEC, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wohlfahrt P, Jenca D, Melenovsky V, Mrazkova J, Sramko M, Kotrc M, Zelizko M, Adamkova V, Lopez-Jimenez F, Pitha J, Kautzner J. Remote, Smart Device-Based Cardiac Rehabilitation After Myocardial Infarction: A Pilot, Randomized Cross-Over SmartRehab Study. Mayo Clin Proc Digit Health. 2024 Jun 20;2(3):352-360. doi: 10.1016/j.mcpdig.2024.06.001. eCollection 2024 Sep. PMID 40206122